CLINICAL TRIAL: NCT01900782
Title: A Randomized, Double-blind, Double-dummy, Multicenter Study of Subcutaneous Secukinumab to Demonstrate Efficacy After Twelve Weeks of Treatment, Compared to Placebo and Etanercept, and to Assess the Safety, Tolerability and Long-term Efficacy up to One Year in Subjects With Moderate to Severe Chronic Plaque-type Psoriasis.
Brief Title: Efficacy and Safety Study of Subcutaneous Secukinumab in Treatment of Subjects With Moderate to Severe Chronic Plaque-type Psoriasis as Compared to Etanercept and Placebo.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAIN457A2314; 2013-000463-83 (EudraCT Number)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dosing Regimen 1 (Experimental): Subcutaneous injection
  Interventions: Biological: Intervention A
- Active Comparator (Active Comparator): Subcutaneous injection
  Interventions: Biological: Intervention B
- Placebo (Placebo Comparator): Subcutaneous injection
  Interventions: Biological: Placebo
- Dosing Regimen 2 (Experimental): Subcutaneous injection
  Interventions: Biological: Intervention A

INTERVENTIONS:
Biological: Intervention A — Prefilled syringe.
  Arms: Dosing Regimen 1; Dosing Regimen 2
Biological: Intervention B — Prefilled syringe.
  Arms: Active Comparator
Biological: Placebo — Prefilled syringe to match experimental drug and active comparator.
  Arms: Placebo

SUMMARY:
This withdrawn study was to assess the safety and efficacy of secukinumab compared to etanercept and placebo in patients who have moderate to severe, chronic, plaque-type psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic plaque-type psoriasis, moderate to severe
* Candidate for systemic therapy defined as having psoriasis not adequately controlled by: topical treatment, phototherapy and/or previous systemic therapy

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque-type
* Ongoing use of treatments not allowed for psoriasis

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
PASI (psoriasis area and severity index) and IGA (investigator's global assessment) | Week 12

SECONDARY OUTCOMES:
PASI (psoriasis area and severity index) and IGA (investigator's global assessment) | Week 52
Vital signs, laboratory values, electrocardiograms (ECG), adverse events | Week 12 and 52
Patient reported outcome questionnaires | Week 12 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals